CLINICAL TRIAL: NCT06785831
Title: Opportunities for Increasing Consumption of Local Fruits and Vegetables in Slovenian Population (NutriPlant)
Brief Title: NutriPlant - Opportunities for Increasing Consumption of Local Fruits and Vegetables
Acronym: NutriPlant
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: University Medical Centre Ljubljana (Other); University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KME 0120-242/2024-2711-4; L7-50154 (Other Grant/Funding Number: Slovenian Research And Innovation Agency); L7-50154 (Other Grant/Funding Number: Ministry of Agriculture, Forestry and Food (Slovenia))
Record Dates: First submitted 2024-12-13; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Functional Constipation; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Psyllium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Intervention include consumption of specific foods, therefore masking to participant and investigatior is not possible. Collected data will be masked for accessor of outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Psyllium (Active Comparator): Psyllium containing 3 g dietary fibre, daily, for 4 weeks
  Interventions: Other: Psyllium
- Sauerkraut (Experimental): Sauerkraut containing 3 g dietary fibre, daily, for 4 weeks
  Interventions: Other: Sauerkraut
- Fresh apples (Experimental): Fresh apples containing 3 g dietary fibre, daily, for 4 weeks
  Interventions: Other: Fresh apples
- Dried apples (Experimental): Dried apples containing 3 g dietary fibre, daily, for 4 weeks
  Interventions: Other: Dried apples

INTERVENTIONS:
Other: Psyllium — Participants will once daily consume predefined amount of psyllium, corresponding to 3 g of dietary fibre, for 28 days.
  Arms: Psyllium
Other: Sauerkraut — Participants will once daily consume predefined amount of sauerkraut, corresponding to 3 g of dietary fibre, for 28 days.
  Arms: Sauerkraut
Other: Fresh apples — Participants will once daily consume predefined amount of fresh apples, corresponding to 3 g of dietary fibre, for 28 days.
  Arms: Fresh apples
Other: Dried apples — Participants will once daily consume predefined amount of dried apples, corresponding to 3 g of dietary fibre, for 28 days.
  Arms: Dried apples

SUMMARY:
The effects of different foods to normal bowel function in adult population will be investigated. A randomised controlled intervention trial will be conducted on about 120 (30 per group) adult (18-70 years) subjects with functional constipation and irritable bowel syndrome with constipation according to the IV. Rome criteria. At least one week before inclusion in the study, patients will stop taking laxatives and other anti-constipation medications. Subjects will be randomly selected to consume one of the test foods (fresh apples, dried apples, sauerkraut) or the active control (psyllium) in the equivalent amount of 3 g of fiber per day for 4 weeks. Subjects will be asked not to change their lifestyle habits, such as diet and physical activity level, and not to take oral laxatives during the period of participation in the study.

ELIGIBILITY:
1. Inclusion criteria:

   * Signed informed consent of the participant to participate in the study
   * Age between 18 and 70 years
   * Functional constipation or irritable bowel syndrome
   * Expressed willingness to eat the investigated food daily (sauerkraut, apples, dried apples or psyllium; period of four weeks)
2. Exclusion criteria:

   * Known allergy to the investigated foods (fresh apples, dried apples, sauerkraut or psyllium)
   * Pregnancy or breastfeeding
   * Previous gastrointestinal surgery with the exception of cholecystectomy and appendectomy
   * Other gastrointestinal diseases (chronic inflammatory bowel disease, celiac disease, gastroparesis, etc.)
   * Serious chronic diseases
   * Introduction of extensive changes in diet or physical activity in the last 4 weeks before the inclusion examination
   * Regular use of laxatives or inability to stop using laxatives for the duration of the study
   * Concurrent participation in another study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of complete spontaneous bowel movements (CSBM) / week | fourth week vs pre-intervention
  Daily measurement of number of complete spontaneous bowel movements

OTHER OUTCOMES:
Change in constipation symptom score (CSC) | fourth week vs pre-intervention
  Measurement with constipation symptom score (0-48 points, higher SCS score mean more severe symptoms)
Change in stool consistency using Bristol stool form (BSF) scale | fourth week vs pre-intervention
  Measurement with Bristol stool form (BSF) scale (Type 1: Separate hard lumps, like nuts (difficult to pass), Type 2: Sausage-shaped, but lumpy, Type 3: Like a sausage but with cracks on its surface, Type 4: Like a sausage or snake, smooth and soft (average stool), Type 5: Soft blobs with clear cut edges, Type 6: Fluffy pieces with ragged edges, a mushy stool (diarrhea), Type 7: Watery, no solid pieces, entirely liquid (diarrhea))
Change in blood lipids | in week after intervention vs pre-intervention
  Laboratory measuremnt of S-Cholesterol, S-HDL-Cholesterol, S-LDL-Cholesterol and S-Triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kušar, PhD, Study Director — Researcher
Locations (1):
- UKC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided